CLINICAL TRIAL: NCT01709838
Title: An Open Label, Multi-center, Efficacy and Safety Study of Deferasirox in Iron Overloaded Patients With Non-transfusion Dependent Thalassemia
Brief Title: Efficacy and Safety Study of Deferasirox in Patients With Non-transfusion Dependent Thalassemia
Acronym: THETIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670E2419; 2012-000650-64 (EudraCT Number)
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Non-transfusion Dependent Thalassemia
Keywords: Non-transfusion dependent thalassemia; NTDT; deferasirox; ICL670; LIC; Liver Iron Concentration
MeSH Terms: interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deferasirox (Other): All patients were treated with 10mg/kg/day deferasirox with dose adjustments after 4 weeks of treatment according to baseline Liver Iron Concentration (LIC).
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox — Deferasirox dispersible tablets at strengths of 125 mg, 250 mg, and 500 mg were administered by oral daily dosing.
  Other Names: ICL670

SUMMARY:
Assessed the efficacy of deferasirox in patients with non-transfusion dependent thalassemia based on change in liver iron concentration from baseline after 52 weeks of treatment. Provided further assessment of the long-term efficacy and safety of deferasirox in NTDT patients with iron overload (LIC ≥ 5 mg Fe/g liver dw and SF ≥ 300 ng/mL) for up to 260 weeks.

ELIGIBILITY:
Inclusion Criteria:

Non-transfusion dependent congenital or chronic anemia inclusive of beta-thalassemia intermedia, HbE beta-thalassemia or alpha-thalassemia intermedia (HbH disease)/ Liver iron concentration >/= 5 mg Fe/g dw Serum Ferritin >/= 300 ng/mL

Exclusion Criteria:

HbS-beta Thalassemia, anticipated regular transfusion program during the study, blood transfusion 6 months prior to study start, significant proteinuria, creatinine clearance </= 40 ml/min, serum creatinine > ULN, ALT >5 x ULN, active hepatitis B or C, cirrhosis

Pediatrics Only:

A patient's weight of at least 20 kg is required to allow dosing of 5 mg/kg with one tablet of 125 mg

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2015-01-03 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Novartis Investigative Site, Nanning, Guangxi, China
- Novartis Investigative Site, Goudi-Athens, GR, Greece
- Italy (2):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Milan, MI
- Novartis Investigative Site, Hazmiyeh, Beyrouth, Lebanon
- Novartis Investigative Site, Bangkok, Thailand
- Novartis Investigative Site, Tunis, Tunisia
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At least 117 patients were planned to be enrolled; 134 patients were enrolled.
Pre-assignment Details: At least 117 patients were planned to be enrolled; 134 patients were enrolled.
Period: Overall Study
Arm/Group | Deferasirox
Started | 134
Completed | 67
Not Completed | 67
Not completed — Withdrawal by Subject | 21
Not completed — Lost to Follow-up | 16
Not completed — Pregnancy | 10
Not completed — Subject/guardian decision | 8
Not completed — Adverse Event | 4
Not completed — Physician Decision | 4
Not completed — Death | 3
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (11.10)
Age, Customized [Number; unit: participants]
  < 18 years | 25
  18 - < 50 years | 104
  50 - < 65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 76
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 85
  Caucasian | 48
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Liver Iron Content (LIC) at 52 Weeks From Baseline
Description: Absolute change in liver iron concentration measured by MRI from baseline after 52 weeks of treatment
Time Frame: Baseline, 52 weeks
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
mg Fe/g dw | -6.68 (7.018)

2. Secondary Outcome: Percentage of Participants With Baseline LIC>15 Achieving LIC<5 mg Fe/g dw
Description: The percentage of participants with baseline LIC>15 mg Fe/g dw achieving an LIC <5 mg Fe/g dw during the study
Time Frame: 5 years
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
percentage of participants | 51.0

3. Secondary Outcome: Time to Achieving LIC <5 mg Fe/g dw
Description: Time to achieving LIC <5 mg Fe/g dw for participants with baseline LIC>15 mg Fe/g dw during the study
Time Frame: 5 years
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
months | 36.3 [28.55 to 48.30]

4. Secondary Outcome: Time From Target LIC of 3 mg Fe/g dw to the First LIC ≥5 mg Fe/g dw in the Follow up Period
Description: Time from the target LIC <3 mg Fe/g dw to the first LIC ≥5 mg Fe/g dw in the follow-up period
Time Frame: post-baseline, up to 260 weeks
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
days | 27.4 [17.68 to NA] — N/A = Not estimable as data is not sufficient to estimate the upper limit

5. Secondary Outcome: Absolute Change in Health-related Outcomes Using Medical Outcomes Study Form 36 (SF-36v2)
Description: The SF-36 is a self-administered questionnaire for adults (from 18 years of age) and contains 36 items which measure: Physical functioning, Role limitation due to physical health problems, Bodily pain, General health perceptions, Vitality, Social functioning, Role limitations due to emotional problems and General mental health . The higher values indicate a better evaluation of health. Range: 0 to 100 [0 (worst possible health state measured by the questionnaire) to 100 (best possible health state)].
Time Frame: Baseline, 52, 104 & 156 Weeks
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Deferasirox
Number analyzed (Participants) | 105
scores on a scale
  Physical Functioning Week 52: number analyzed (Participants) | 89
  Physical Functioning Week 52 | -0.5 (5.5)
  Physical Functioning Week 104: number analyzed (Participants) | 74
  Physical Functioning Week 104 | -0.7 (4.9)
  Physical Functioning Week 156: number analyzed (Participants) | 64
  Physical Functioning Week 156 | 0.6 (6.1)
  Role Physical Week 52: number analyzed (Participants) | 89
  Role Physical Week 52 | 0.9 (9.1)
  Role Physical Week 104: number analyzed (Participants) | 74
  Role Physical Week 104 | -1.0 (10.2)
  Role Physical Week 156: number analyzed (Participants) | 64
  Role Physical Week 156 | 1.0 (10.9)
  Bodily Pain Week 52: number analyzed (Participants) | 89
  Bodily Pain Week 52 | -0.0 (11.6)
  Bodily Pain Week 104: number analyzed (Participants) | 74
  Bodily Pain Week 104 | -1.3 (10.8)
  General Health Week 52: number analyzed (Participants) | 89
  General Health Week 52 | -2.3 (9.1)
  Bodily Pain Week 156: number analyzed (Participants) | 64
  Bodily Pain Week 156 | 0.9 (12.2)
  General Health Pain Week 104: number analyzed (Participants) | 74
  General Health Pain Week 104 | -1.9 (9.2)
  General Health Week 156: number analyzed (Participants) | 64
  General Health Week 156 | -1.1 (8.6)
  Vitality Week 52: number analyzed (Participants) | 89
  Vitality Week 52 | 1.1 (9.7)
  Vitality Week 104: number analyzed (Participants) | 74
  Vitality Week 104 | -0.2 (8.7)
  Vitality Week 156: number analyzed (Participants) | 64
  Vitality Week 156 | 2.1 (9.6)
  Social Functioning Week 52: number analyzed (Participants) | 89
  Social Functioning Week 52 | 0.9 (9.8)
  Social Functioning Week 104: number analyzed (Participants) | 74
  Social Functioning Week 104 | -1.2 (9.6)
  Social Functioning Week 156: number analyzed (Participants) | 64
  Social Functioning Week 156 | 1.6 (10.6)
  Role Emotional Week 52: number analyzed (Participants) | 89
  Role Emotional Week 52 | -0.1 (11.3)
  Role Emotional Week 104: number analyzed (Participants) | 74
  Role Emotional Week 104 | -2.5 (12.2)
  Role Emotional Week 156: number analyzed (Participants) | 64
  Role Emotional Week 156 | 0.7 (11.2)
  Mental Health Week 52: number analyzed (Participants) | 88
  Mental Health Week 52 | 1.5 (11.7)
  Mental Health Week 104: number analyzed (Participants) | 73
  Mental Health Week 104 | -0.6 (11.4)
  Mental Health Week 156: number analyzed (Participants) | 63
  Mental Health Week 156 | 2.8 (10.9)
  Physical Component Week 52: number analyzed (Participants) | 89
  Physical Component Week 52 | -0.8 (7.2)
  Physical Component Week 104: number analyzed (Participants) | 74
  Physical Component Week 104 | -1.0 (7.4)
  Physical Component Week 156: number analyzed (Participants) | 64
  Physical Component Week 156 | -0.1 (7.9)
  Mental Component Week 104: number analyzed (Participants) | 73
  Mental Component Week 104 | -1.3 (11.1)
  Mental Component Week 52: number analyzed (Participants) | 88
  Mental Component Week 52 | 1.1 (10.9)
  Mental Component Week 156: number analyzed (Participants) | 63
  Mental Component Week 156 | 2.2 (10.8)
  SF6D Health Utility Index Week 52: number analyzed (Participants) | 88
  SF6D Health Utility Index Week 52 | 0.0 (0.1)
  SF6D Health Utility Index Week 104: number analyzed (Participants) | 73
  SF6D Health Utility Index Week 104 | -0.0 (0.1)
  SF6D Health Utility Index Week 156: number analyzed (Participants) | 63
  SF6D Health Utility Index Week 156 | 0.0 (0.1)

6. Secondary Outcome: Absolute Change in Health-related Outcomes Using the Pediatric Quality of Life Questionnaire (PedsQL™)
Description: The PedsQL™ is a modular approach to measuring health-related quality of life (HRQOL) in children and adolescents. The 23-item PedsQL™ Generic Core Scales encompass the essential core domains for pediatric HRQOL measurement: 1) Physical Functioning (8 items), 2) Emotional Functioning (5 items), 3) Social Functioning (5 items), and 4) School Functioning (5 items). The Generic Core Scales are designed to enable comparisons across patient and healthy populations. The higher values indicate a better evaluation of health. Range: 0 to 100 [0 (worst possible health state measured by the questionnaire) to 100 (best possible health state)].
Time Frame: Baseline, 52, 104 & 156 Weeks
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Deferasirox
Number analyzed (Participants) | 16
scores on a scale
  Physical Functioning - Teenager Wk 52: number analyzed (Participants) | 15
  Physical Functioning - Teenager Wk 52 | 2.3 (13.7)
  Physical Functioning - Teenager Wk 104: number analyzed (Participants) | 13
  Physical Functioning - Teenager Wk 104 | 1.0 (19.3)
  Physical Functioning - Teenager Wk 156: number analyzed (Participants) | 11
  Physical Functioning - Teenager Wk 156 | -0.9 (15.4)
  Emotional Functioning - Teenager Wk 52: number analyzed (Participants) | 15
  Emotional Functioning - Teenager Wk 52 | 0.7 (17.8)
  Emotional Functioning - Teenager Wk 104: number analyzed (Participants) | 13
  Emotional Functioning - Teenager Wk 104 | 3.1 (27.6)
  Emotional Functioning - Teenager Wk 156: number analyzed (Participants) | 11
  Emotional Functioning - Teenager Wk 156 | 10.9 (25.9)
  Social Functioning - Teenager Wk 52: number analyzed (Participants) | 15
  Social Functioning - Teenager Wk 52 | -9.3 (17.5)
  Social Functioning - Teenager Wk 104: number analyzed (Participants) | 13
  Social Functioning - Teenager Wk 104 | -10.0 (17.8)
  Social Functioning - Teenager Wk 156: number analyzed (Participants) | 11
  Social Functioning - Teenager Wk 156 | -5.0 (20.1)
  School Functioning - Teenager Wk 52: number analyzed (Participants) | 14
  School Functioning - Teenager Wk 52 | 0.7 (12.4)
  School Functioning - Teenager Wk 104: number analyzed (Participants) | 12
  School Functioning - Teenager Wk 104 | -3.8 (16.4)
  School Functioning - Teenager Wk 156: number analyzed (Participants) | 10
  School Functioning - Teenager Wk 156 | 1.0 (21.4)
  Physical Health - Teenager Wk 52: number analyzed (Participants) | 15
  Physical Health - Teenager Wk 52 | 2.3 (13.7)
  Physical Health - Teenager Wk 104: number analyzed (Participants) | 13
  Physical Health - Teenager Wk 104 | 1.0 (19.3)
  Physical Health - Teenager Wk 156: number analyzed (Participants) | 11
  Physical Health - Teenager Wk 156 | -0.9 (15.4)
  Psychosocial Health - Teenager Wk 52: number analyzed (Participants) | 15
  Psychosocial Health - Teenager Wk 52 | -3.3 (13.0)
  Psychosocial Health - Teenager Wk 104: number analyzed (Participants) | 13
  Psychosocial Health - Teenager Wk 104 | -4.0 (16.9)
  Psycholosocial Health - Teenager Wk 156: number analyzed (Participants) | 11
  Psycholosocial Health - Teenager Wk 156 | 2.0 (19.1)
  Total Score - Teenager Wk 52: number analyzed (Participants) | 15
  Total Score - Teenager Wk 52 | -1.0 (10.6)
  Total Score - Teenager Wk 104: number analyzed (Participants) | 13
  Total Score - Teenager Wk 104 | -1.9 (14.4)
  Total Score - Teenager Wk 156: number analyzed (Participants) | 11
  Total Score - Teenager Wk 156 | 1.2 (15.8)
  Physical Functioning - Parent Wk 52: number analyzed (Participants) | 15
  Physical Functioning - Parent Wk 52 | -2.9 (19.0)
  Physical Functioning - Parent Wk 104: number analyzed (Participants) | 13
  Physical Functioning - Parent Wk 104 | 0.0 (18.6)
  Physical Functioning - Parent Wk 156: number analyzed (Participants) | 10
  Physical Functioning - Parent Wk 156 | -0.3 (15.6)
  Emotional Functioning - Parent Wk 52: number analyzed (Participants) | 15
  Emotional Functioning - Parent Wk 52 | -8.7 (19.1)
  Emotional Functioning - Parent Wk 104: number analyzed (Participants) | 13
  Emotional Functioning - Parent Wk 104 | -3.8 (20.8)
  Emotional Functioning - Parent Wk 156: number analyzed (Participants) | 10
  Emotional Functioning - Parent Wk 156 | 2.0 (20.6)
  Social Functioning - Parent Wk 52: number analyzed (Participants) | 15
  Social Functioning - Parent Wk 52 | -3.7 (15.5)
  Social Functioning - Parent Wk 104: number analyzed (Participants) | 13
  Social Functioning - Parent Wk 104 | -4.6 (18.0)
  Social Functioning - Parent Wk 156: number analyzed (Participants) | 10
  Social Functioning - Parent Wk 156 | -6.0 (20.9)
  School Functioning - Parent Wk 52: number analyzed (Participants) | 14
  School Functioning - Parent Wk 52 | -3.6 (20.6)
  School Functioning - Parent Wk 104: number analyzed (Participants) | 12
  School Functioning - Parent Wk 104 | 0.0 (11.7)
  School Functioning - Parent Wk 156: number analyzed (Participants) | 9
  School Functioning - Parent Wk 156 | -0.6 (21.1)
  Physical Health - Parent Wk 52: number analyzed (Participants) | 15
  Physical Health - Parent Wk 52 | -2.9 (19.0)
  Physical Health - Parent Wk 104: number analyzed (Participants) | 13
  Physical Health - Parent Wk 104 | 0.0 (18.6)
  Physical Health - Parent Wk 156: number analyzed (Participants) | 10
  Physical Health - Parent Wk 156 | -0.3 (15.6)
  Psychosocial Health - Parent Wk 52: number analyzed (Participants) | 15
  Psychosocial Health - Parent Wk 52 | -5.5 (15.0)
  Psychosocial Health - Parent Wk 104: number analyzed (Participants) | 13
  Psychosocial Health - Parent Wk 104 | -3.2 (12.3)
  Psychosocial Health - Parent Wk 156: number analyzed (Participants) | 10
  Psychosocial Health - Parent Wk 156 | -1.8 (14.1)
  Total Score - Parent Wk 52: number analyzed (Participants) | 15
  Total Score - Parent Wk 52 | -4.6 (14.8)
  Total Score - Parent Wk 104: number analyzed (Participants) | 13
  Total Score - Parent Wk 104 | -1.9 (12.0)
  Total Score - Parent Wk 156: number analyzed (Participants) | 10
  Total Score - Parent Wk 156 | -1.1 (12.9)

7. Secondary Outcome: Absolute Change in LIC From Baseline Over Time
Description: Absolute change in serum ferritin from baseline over time up to 260 weeks
Time Frame: 24, 52, 76, 104, 128, 156, 180, 208, 232, 260 Weeks
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
mg Fe/g dw
  Week 24: number analyzed (Participants) | 126
  Week 24 | -3.67 (3.778)
  Week 52: number analyzed (Participants) | 118
  Week 52 | -7.02 (7.132)
  Week 76: number analyzed (Participants) | 107
  Week 76 | -8.93 (8.922)
  Week 104: number analyzed (Participants) | 100
  Week 104 | -9.63 (9.474)
  Week 128: number analyzed (Participants) | 95
  Week 128 | -10.03 (9.445)
  Week 156: number analyzed (Participants) | 92
  Week 156 | -10.20 (9.746)
  Week 180: number analyzed (Participants) | 86
  Week 180 | -9.94 (9.838)
  Week 208: number analyzed (Participants) | 81
  Week 208 | -10.04 (10.010)
  Week 232: number analyzed (Participants) | 66
  Week 232 | -10.58 (10.045)
  Week 260: number analyzed (Participants) | 66
  Week 260 | -10.57 (10.366)

8. Secondary Outcome: Serum Ferritin (SF) vs LIC at Baseline and EOS (Week 260 + 30 Days Follow-up)
Description: Correlation between serum ferritin and LIC is assessed using scatter plots with pearson correlation coefficient and simple linear model.
Time Frame: Baseline, End of Study (EOS): Week 260 + 30 days follow up
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Number; unit: correlation coefficient
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
correlation coefficient
  At Baseline | 0.730
  Change from Baseline at EOS: number analyzed (Participants) | 77
  Change from Baseline at EOS | 0.531

9. Secondary Outcome: Correlation Analysis for Absolute Change in LIC and Serum Ferritin at Week 24 and EOS (Week 260 + 30 Days Follow-up)
Description: Correlation for absolute change between LIC and serum ferritin was assessed using scatter plots with pearson correlation coefficient and simple linear model.
Time Frame: Week 24, End of Study (EOS): Week 260 + 30 days follow up
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Number; unit: correlation coefficient
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
correlation coefficient
  Week 24: number analyzed (Participants) | 125
  Week 24 | 0.299
  Change from Baseline at EOS: number analyzed (Participants) | 77
  Change from Baseline at EOS | 0.740

10. Secondary Outcome: Absolute Change in LIC From Baseline After 52 Weeks of Treatment by Underlying Non-transfusion Dependent Thalassemia (NTDT) Syndrome
Description: Absolute change in liver iron concentration measured by MRI from baseline after 52 weeks of treatment by underlying NTDT syndrome. The 4 underlying disease types: Beta-thalassemia intermedia (N =69), HbE beta-thalassemia (N = 24), Alpha-thalassemia intermedia (HbH disease) (N = 40), Other, specify (N = 1)
Time Frame: Baseline, 52 Weeks
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
mg Fe/g dw
  Beta-thalassemia intermedia: number analyzed (Participants) | 65
  Beta-thalassemia intermedia | -6.11 (6.481)
  HbE beta-thalassemia: number analyzed (Participants) | 23
  HbE beta-thalassemia | -6.18 (7.572)
  Alpha-thalassemia intermedia (HbH disease): number analyzed (Participants) | 38
  Alpha-thalassemia intermedia (HbH disease) | -7.97 (7.652)
  Other, specify: number analyzed (Participants) | 1
  Other, specify | -6.00 (NA) — N/A: Standard Deviation cannot be obtained for 1 patient

11. Secondary Outcome: Absolute Change in Serum Ferritin From Baseline After 52 Weeks
Description: Absolute change in serum ferritin from baseline after 52 weeks of treatment
Time Frame: Baseline, 52 weeks
Population: The Full Analysis Set (FAS) consisted of all patients who were assigned at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Deferasirox
Number analyzed (Participants) | 134
ng/mL | -494.64 (760.782)

12. Secondary Outcome: PK Parameters: AUCtau
Description: The pharmacokinetic parameter, AUCtau was determined using non-compartmental method(s) for deferasirox and its iron complex. AUC=area under the concentration-time curve during a dosing interval at steady state (amount × time × volume).
Time Frame: pre-dose (0 hour), and at 2, and 4 hours at Week 4
Population: The PK analysis set consisted of all patients from FAS who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*umol/L
Arm/Group | Deferasirox
Number analyzed (Participants) | 22
hr*umol/L | 678.2 (61.9)

13. Secondary Outcome: PK Parameters: Cmax
Description: The pharmacokinetic parameter, Cmax, was determined using non-compartmental method(s) for deferasirox and its iron complex. Cmax (maximum/peak plasma drug concentration after drug administration)=amount × volume
Time Frame: pre-dose (0 hour), and at 2, and 4 hours at Week 4
Population: The PK analysis set consisted of all patients from FAS who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: umol/L
Arm/Group | Deferasirox
Number analyzed (Participants) | 22
umol/L | 53.367 (60.960)

14. Secondary Outcome: PK Parameters: Tmax
Description: The pharmacokinetic parameter, Tmax, may be determined using non-compartmental method(s) for deferasirox and its iron complex. Tmax=time to reach maximum/peak concentration following drug administration.
Time Frame: pre-dose (0 hour), and at 2, and 4 hours at Week 4
Population: The PK analysis set consisted of all patients from FAS who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Deferasirox
Number analyzed (Participants) | 22
hr | 2.5131 (33.9321)

15. Secondary Outcome: Plasma Pharmacokinetics (PK) Deferasirox Concentrations
Description: Blood samples for PK evaluation were collected for a sub-group of patients. The patient had to have been on treatment without dose adjustment or treatment interruption (for any reason) for at least 4 consecutive days prior to scheduled PK sampling visit. If there was a dosage change or interruption within 4 days of the visit, no PK blood samples was collected, and an appropriate comment had to be made on the PK CRF page.
Time Frame: Weeks 12 & 24: pre-dose (0hr), 2hr & 4hr post-dose
Population: The PK analysis set consisted of all patients from FAS who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*umol/L
Arm/Group | Deferasirox
Number analyzed (Participants) | 22
hr*umol/L
  4 weeks: 0hr pre-dose | 6.513 (75.891)
  4 weeks: 2hr post-dose | 48.556 (58.006)
  4 weeks: 4hr post-dose | 44.652 (69.392)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 63.2 months.
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 7 years.
Groups:
- Chinese: This group was comprised of Chinese participants only
- Non-Chinese: This group was comprised of non- Chinese participants only
- All Patients: This group was comprised of all patients: Chinese and non-Chinese participants
Arm/Group | Chinese | Non-Chinese | All Patients
All-Cause Mortality (participants affected / at risk) | 2/68 | 0/66 | 2/134
Serious Adverse Events (participants affected / at risk) | 15/68 | 30/66 | 45/134
Other Adverse Events (participants affected / at risk) | 26/68 | 58/66 | 84/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chinese (N=68) | Non-Chinese (N=66) | All Patients (N=134)
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 6
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 0 | 2 | 2
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Hypersplenism (Blood and lymphatic system disorders) | 2 | 0 | 2
Splenomegaly (Blood and lymphatic system disorders) | 2 | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 2 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Superior mesenteric artery syndrome (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 0 | 2 | 2
Generalised oedema (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 3 | 3
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 3 | 4
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 2
Epididymitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 4 | 4
Lung infection (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 2
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 3 | 4 | 7
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 3
Varicella (Infections and infestations) | 0 | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chinese (N=68) | Non-Chinese (N=66) | All Patients (N=134)
Anaemia (Blood and lymphatic system disorders) | 0 | 5 | 5
Abdominal discomfort (Gastrointestinal disorders) | 2 | 5 | 7
Abdominal pain (Gastrointestinal disorders) | 0 | 15 | 15
Abdominal pain upper (Gastrointestinal disorders) | 0 | 9 | 9
Constipation (Gastrointestinal disorders) | 0 | 4 | 4
Dental caries (Gastrointestinal disorders) | 0 | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 19 | 20
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 4
Gastritis (Gastrointestinal disorders) | 0 | 5 | 5
Nausea (Gastrointestinal disorders) | 2 | 10 | 12
Toothache (Gastrointestinal disorders) | 0 | 7 | 7
Vomiting (Gastrointestinal disorders) | 1 | 11 | 12
Fatigue (General disorders) | 1 | 12 | 13
Influenza like illness (General disorders) | 0 | 7 | 7
Pyrexia (General disorders) | 3 | 14 | 17
Cholelithiasis (Hepatobiliary disorders) | 1 | 6 | 7
Conjunctivitis (Infections and infestations) | 0 | 5 | 5
Gastroenteritis (Infections and infestations) | 1 | 9 | 10
Influenza (Infections and infestations) | 0 | 11 | 11
Pharyngitis (Infections and infestations) | 0 | 11 | 11
Tonsillitis (Infections and infestations) | 0 | 12 | 12
Upper respiratory tract infection (Infections and infestations) | 7 | 27 | 34
Urinary tract infection (Infections and infestations) | 2 | 8 | 10
Blood creatinine increased (Investigations) | 1 | 4 | 5
Platelet count increased (Investigations) | 13 | 1 | 14
Urine protein/creatinine ratio increased (Investigations) | 0 | 6 | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 8 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 5 | 6
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 8 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 16 | 16
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 10 | 10
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 6
Dizziness (Nervous system disorders) | 0 | 8 | 8
Headache (Nervous system disorders) | 0 | 27 | 27
Anxiety (Psychiatric disorders) | 0 | 4 | 4
Insomnia (Psychiatric disorders) | 0 | 5 | 5
Dysuria (Renal and urinary disorders) | 0 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 16 | 16
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 8
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT01709838/SAP_000.pdf
  • Study Protocol (2014-09-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT01709838/Prot_001.pdf